# Written Language Intervention for Functional Texts (WLIFT) Consent Form

**Baylor University** 

#### **Communication Sciences and Disorders**

Consent Form for Research

PROTOCOL TITLE: Written Language Intervention for Functional Texts for Young Adults with

Intellectual and Developmental Disabilities

PRINCIPAL INVESTIGATOR: Alison Prahl, PhD, CCC-SLP

Last Updated: 04/20/2023

#### Important Information about this Research Study

I am a professor and speech-language pathologist from Baylor University in Waco, TX. We are doing a research study about teaching strategies to help you understand the things that you read daily, such as text messages, social media, or emails. We would like your help. You do not have to do this if you do not want to. If you say yes now, you can still stop at any time. Feel free to ask if you do not understand anything in this form.

### What will happen if I take part in this research study?

If you want to, you will meet with a member of the research team for an initial study visit on a video call on the computer using Zoom to make sure the study is a good fit for you. If it is a good fit, you

will complete Sessions 1 and 2 (scheduled 3 months apart) on Zoom which will include some reading activities. Lastly, Session 3 also includes reading activities and will be scheduled 6 months later.

You will also be assigned by chance (like a coin toss) to one of two study groups. One group will be the control group who will receive their reading activity results and tips to support their reading at the conclusion of the study. The other group will be the treatment group who will meet with a member of the research team two times each week for about 45-minutes via teletherapy. You and the researcher cannot choose your study group. You will have an equal chance of being assigned to either study group.

For the treatment group, your education, community program staff, or family will help schedule the sessions and make sure you have access to the teletherapy sessions, as well as make sure you have any other materials you may need. During the teletherapy sessions, the research team member will teach you strategies to help you understand the things that you read daily, such as text messages, social media, or emails. The research team member will show you how to use the strategies, then you all will practice together, then you will practice on your own when you are ready. If needed, the research team member will be with you on the computer to help you. Because the strategies are for reading things like messages and emails, we may ask you to share your reading materials (e.g., text messages, emails) with the research team towards the end of the study. At the end of the study, you will be asked to complete a short survey and we will ask you what you liked and did not like about the strategies.

If you say yes, you will be in the research study for about nine months. About 50 young adults will take part in this research study.

#### What are the risks of taking part in this research study?

If you would like to stop at any time for any reason, just tell Dr. Alison Prahl. It will not be a problem. It is your choice if you want to stop at any time. If you decide that you want to stop across three sessions in a row, we will talk to you to see if you would like to end the study.

#### Are there any benefits from being in this research study?

If you say yes, you will help give us information about strategies that help students in programs like yours to read successfully. We will not share your name in our findings or with anyone except the people who work on this research project.

#### **How Will You Protect my Information?**

A risk of taking part in this study is the possibility of a loss of confidentiality. Loss of confidentiality includes having your personal information shared with someone who is not on the study team and was not supposed to see or know about your information. The researcher plans to protect your confidentiality.

We will be recording the sessions for our study so that we remember what you say and how the research team member teaches you the strategies. Only members of the research team will know what you say. Recordings will be stored for up to five years. We will not use your real name or the names of anyone else you mention. We will destroy this document and any data about you five years after the results of the study are published. Until then, we will keep all information locked in a file cabinet in Dr. Prahl's lab and all electronic data stored on a secure server at Baylor University.

A description of this study will be available on http://www.ClinicalTrials.gov as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## Will information you collect about me be used for future research studies?

Information collected from you as part of this research may be shared with the research community. We will not share your name in or findings with anyone except the people who work on this research project.

#### Will I be compensated for being part of the study?

You will receive up to \$225.00 in your choice of either payment cards or electronic Amazon gift cards for your time over the nine-month study. The payment schedule is as follows. Once you complete the screening visit, you will receive \$25. Once you complete the Session 1 visit, you will receive \$50. Once you complete the Session 2 visit, you will receive \$75. Once you complete the Session 3 visit, you will receive \$75. If you are randomly assigned to the control group, you will receive \$50 after the study is completed. If you complete the entire screening visit, but are not eligible to participate in the study, you will receive a \$25.00 payment card or electronic Amazon gift card.

Per University Policy, to pay you we will need to collect your social security number or Individual Taxpayer Identification Number for tax purposes. If you do not want to provide this information, you can still be in the research study, but we cannot pay you.

Is it possible that I will be asked to leave the study?

The researcher may take you out of this study without your permission. This may happen because the researcher thinks it is in your best interest or you can't make the required study visits.

#### **Your Participation in this Study is Voluntary**

Taking part in this study is your choice. You are free not to take part or to withdraw at any time for any reason. No matter what you decide, there will be no penalty or loss of benefit to which you are entitled. If you decide to withdraw from this study, the information that you have already provided will be kept confidential. You cannot withdraw information collected prior to your withdrawal.

## Contact Information for the Study Team and Questions about the Research

If you have any questions, please contact Dr. Alison Prahl at Baylor University. You can reach me at 254-710-2572 or alison\_prahl@baylor.edu.

If you have questions about your rights as a research participant, or wish to obtain information, ask questions, or discuss any concerns about this study with someone other than the researcher(s), please contact the Baylor University Institutional Review Board, Office of the Vice Provost for Research at 254-710-3708 or irb@baylor.edu.

#### **Your Consent**

By selecting "Yes" below, you are agreeing to be in this study. We will give you a copy of this document for your records and we will keep a copy. If you have any questions about the study after you electronically agree, you can contact the study team using the information provided above.

| I understand what the study is about and my questions so far have been answered. |
|---|
| Please indicate in the survey questions below whether you want to participate. |
| My name: |
| My name: |
| I give my consent to participate in the study. |
| Yes |
| O No |
| I give permission to be audio/video recorded. |
| Yes |
| O No |
| I agree for the research team to use my video recordings in |

teaching or professional development workshops.

| O Yes |
|---|
| O No |
| I give the research team permission to keep my contact |
| information and to contact me for future research projects. |
| O Yes |
| O No |
| Phone number: |
| E-mail address: |
| L THAII Address. |
| NA/less and a second and in action as in the action as in the action of |
| Why are you participating in the research study? |

| What do you hope to get out of this research study? |
|-----------------------------------------------------|

Powered by Qualtrics